CLINICAL TRIAL: NCT01733953
Title: Pilot Study of Statin Therapy in Young Adult Survivors of Childhood Cancer
Brief Title: Statin Therapy in Young Adult Survivors of Childhood Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1207M17202
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Disease; Childhood ALL; Childhood NHL
Keywords: Cardiovascular Disease; Childhood ALL; Childhood NHL
MeSH Terms: conditions — Cardiovascular Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): 6-Months Atorvastatin Therapy; 40mg oral, once daily
  Interventions: Drug: Atorvastatin
- Sugar Pill (Placebo) (Placebo Comparator): 6-Months Placebo (sugar pill); oral, once daily
  Interventions: Drug: Sugar Pill (Placebo)

INTERVENTIONS:
Drug: Atorvastatin — 6-Months of Atorvastatin (Lipitor); 40mg, oral, once daily.
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Sugar Pill (Placebo) — 6-Months of placebo (sugar) pill; oral, once daily
  Other Names: Placebo
  Arms: Sugar Pill (Placebo)

SUMMARY:
Adult survivors of childhood cancer are at high risk of developing cardiovascular disease. Therapies used to treat many cancers, such as chemotherapy and radiation, likely cause damage to the surface of the artery wall called the endothelial layer, leading to the induction of atherosclerosis and eventual cardiovascular disease. HMG coenzyme A reductase inhibitors, or statins, improve endothelial function independent of cholesterol-lowering. In addition, statins have been shown to reduce arterial stiffness and slow arterial thickening. Despite strong evidence supporting the vascular benefits of statins in many different patient populations, these medications have never been studied in cancer survivors. Therefore, the overall objective of this study is to evaluate the effects of statin therapy on vascular health in young adult survivors of childhood cancer.

Twenty-four young adult (age 18-39 years old) survivors of childhood acute lymphoblastic leukemia (ALL) or non-Hodgkin's lymphoma (NHL) will be enrolled in a six-month randomized, double-blind (participants and investigators), placebo-controlled pilot clinical trial comparing the effects of atorvastatin versus placebo on endothelial function and other measures of vascular health.

Our primary objective is to evaluate the effects of 6-months of statin therapy on conduit artery endothelial function in young adult survivors of childhood cancer. The investigators hypothesize that, compared to placebo, atorvastatin will significantly increase brachial artery flow-mediated dilation in survivors of childhood acute lymphoblastic leukemia and non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Adult survivors of childhood cancer are at seven times the risk of dying from cardiovascular disease compared to the general population. The increased risk is thought to be the result of the therapies used to treat the cancer such as chemotherapy and radiation. These therapies likely cause damage to the endothelial cells, which line the arterial wall and, when function properly, offer protection from atherosclerosis. Young adult survivors of childhood ALL have reduced endothelial function, or endothelial dysfunction, compared to healthy controls. Endothelial dysfunction is considered an early manifestation of atherosclerosis and therefore is an ideal target of therapy in order to reduce the risk of cardiovascular disease. Interventions that improve endothelial function in young adult survivors of childhood cancer may be beneficial in terms of mitigating the medium- and long-term risk of developing this chronic disease.

HMG coenzyme A reductase inhibitors, or statins, are widely used for cardiovascular disease risk reduction. These medications are primarily used to reduce levels of total- and low-density lipoprotein (LDL) -cholesterol. Meta-analyses have consistently demonstrated that statin therapy improves endothelial function in a wide array of patient populations. Beyond their well-described vascular benefits, statins are an attractive therapeutic option for cardiovascular disease risk reduction due to their strong safety profile.

Despite the clear potential for endothelial function improvement and cardiovascular risk reduction, statin therapy has never been evaluated in survivors of childhood cancer. Although statins have been well-studied in other patient populations at risk for cardiovascular disease, there is strong justification for evaluation in cancer survivors since the mechanisms responsible for the vascular problems in these individuals (treatment-induced vascular toxicity) differ from traditional atherosclerosis. Therefore, the objective of the current study is to assess the ability of statin therapy to improve endothelial function, arterial stiffness, and arterial thickening in young adult survivors of childhood cancer. The focus of the study will be on survivors of hematologic malignancies, acute lymphoblastic leukemia (ALL) and non-Hodgkin's lymphoma (NHL), since the former has been shown to be associated with endothelial impairments and both cancers share common treatment exposures (chemotherapy and radiation), which is likely the primary factor responsible for endothelial dysfunction in these individuals.

Twenty-four young adult (age 18-39 years old) survivors of childhood acute lymphoblastic leukemia (ALL) and non-Hodgkin's lymphoma (NHL)will be enrolled in a six-month randomized, double-blind (participants and investigators), placebo-controlled pilot clinical trial comparing the effects of atorvastatin versus placebo on endothelial function and other measures of vascular health. Following baseline testing, subjects will be randomly assigned (1:1) to either atorvastatin or placebo. Participants will return at 1-month and 3-months for assessment of safety (blood draw and adverse event assessment) and medication compliance and at 6-months for assessment of safety, medication compliance, and reassessment of baseline variables.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of childhood acute lymphoblastic leukemia (ALL) or non-Hodgkins's lymphoma (NHL) (treated for ALL or NHL before the age of 21 years old and ≥5 years post-treatment)
* 18-39 years old

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Prior treatment with hematopoietic stem cell transplant
* Low-density lipoprotein (LDL) -cholesterol ≥130 mg/dL (individuals with elevated LDL-cholesterol will be referred for clinical management of dyslipidemia)
* Alanine transaminase (ALT), Aspartate transaminase (AST), or Creatine kinase (CK) greater than 2 times the upper limit of normal
* Current or recent (within 6-months) use of lipid-lowering medication
* Recent initiation (within 6-months) of anti-hypertensive medication (individuals on stable therapy may be enrolled)
* Current or recent (within 6-months) use of fibric acid derivatives, lipid-modifying doses of niacin, cyclosporine or strong CYP3A4 inhibitors (i.e. clarithromycin, HIV protease inhibitors, and itraconazole)
* Pregnant, lactating or planning to become pregnant
* Liver/renal dysfunction

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Kelly, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
At this time we have no plan to share the IPD.

REFERENCES:
- [Derived] Marlatt KL, Steinberger J, Rudser KD, Dengel DR, Sadak KT, Lee JL, Blaes AH, Duprez DA, Perkins JL, Ross JA, Kelly AS. The Effect of Atorvastatin on Vascular Function and Structure in Young Adult Survivors of Childhood Cancer: A Randomized, Placebo-Controlled Pilot Clinical Trial. J Adolesc Young Adult Oncol. 2019 Aug;8(4):442-450. doi: 10.1089/jayao.2017.0075. Epub 2017 Aug 30. PMID 28853979

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Started | 14 | 13
Completed | 9 | 6
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Sugar Pill (Placebo) | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (5.7) | 26.9 (6.9) | 26.8 (6.2)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brachial Artery Flow-Mediated Dilation at 6-months
Time Frame: Baseline and 6-Months
Population: Physician withdrawals, loss to follow-up, drug compliance <70%, unrelated injury, and self-withdrawal reduced number analyzed. Also, participant movement during FMD assessment and/or poor ultrasound image quality due to difficult brachial artery anatomy or poor circulation led to some unusable data and thus lowered the analyzable sample size.
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 8 | 3
percentage change | -0.5 [-2.9 to 1.9] | -3.4 [-7.3 to 0.6]

2. Secondary Outcome: Change From Baseline in Carotid Artery Compliance at 6-Months
Description: Carotid Artery Compliance is a measure of arterial stiffness. Higher arterial stiffness places persons at higher risk for CVD.
Time Frame: Baseline and 6-Months
Population: Discrepant sample sizes are due to lack of reliability of measures. If measures were unreliable they were excluded.
Measure: Mean (95% Confidence Interval); unit: mm/mmHg x 10^-3
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 9 | 5
mm/mmHg x 10^-3 | -.34 [-1.4 to 0.7] | 0.57 [-.8 to 2.0]

3. Secondary Outcome: Change From Baseline in Carotid Artery Distensibility at 6-Months
Time Frame: Baseline and 6-Months
Population: Discrepant sample sizes are due to lack of reliability of measures. If measures were unreliable they were excluded.
Measure: Mean (95% Confidence Interval); unit: % distensibility
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 9 | 5
% distensibility | 0.31 [-1.28 to 1.9] | 0.33 [-1.81 to 2.47]

4. Secondary Outcome: Change From Baseline in Pulse Wave Velocity at 6-Months
Time Frame: Baseline and 6-Months
Population: Discrepant sample sizes are due to lack of reliability of measures. If measures were unreliable they were excluded.
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 9 | 5
m/s | -0.52 [-2.06 to 1.02] | -0.3 [-2.36 to 1.76]

5. Secondary Outcome: Change From Baseline in Augmentation Index at 6-Months
Time Frame: Baseline and 6-Months
Population: Discrepant sample sizes are due to lack of reliability of measures. If measures were unreliable they were excluded.
Measure: Mean (95% Confidence Interval); unit: P2/P1
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 9 | 4
P2/P1 | -0.66 [-15.38 to 14.06] | -6.01 [-24.16 to 12.15]

6. Secondary Outcome: Change From Baseline in Carotid Intima-Media Thickness at 6-Months
Time Frame: Baseline and 6-Months
Population: Discrepant sample sizes are due to lack of reliability of measures. If measures were unreliable they were excluded.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Number analyzed (Participants) | 9 | 5
mm | -.01 [-.03 to 0.01] | 0.01 [-0.02 to 0.04]

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Sugar Pill (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No